CLINICAL TRIAL: NCT02725684
Title: Using Genomic Analysis to Guide Individual Treatment in Glioblastoma
Status: Completed | Type: Observational
Sponsor: Rockefeller University (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); Lenox Hill Hospital (Other); North Shore University Hospital (Other); NYU Langone Health (Other); Weill Medical College of Cornell University (Other); Albert Einstein College of Medicine (Other); New York Genome Center (Other)
Responsible Party: Sponsor
Other Study IDs: RDA-0837
Record Dates: First submitted 2015-12-08; First posted 2016-04-01 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Unused samples retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Glioblastoma: Observational study, no intervention
  Interventions: Other: Observational study, no intervention

INTERVENTIONS:
Other: Observational study, no intervention — Observational study, no intervention

SUMMARY:
The purpose of this study is to assess whether the use of genomics can help identify patient specific treatment choices in cancer. In order to test this, the investigators plan to use genomic sequencing technology to identify patient specific mutations in glioblastoma multiforme (GBM) as compared to normal cells to identify mutations. Further analysis will identify potential treatment targets and whether there are any drugs that could be used for these particular mutations. Follow up clinical data will be assessed to see if this individualized method of choosing treatment options can improve clinical outcomes in patients with GBM.

DETAILED DESCRIPTION:
The purpose of the study is to assess whether the use of genomics can identify patient specific treatment choices in glioblastoma (GBM) that improves clinical outcomes over standard of care. GBM is a devastating disease, the most common primary brain tumor and the most aggressive. With current standard therapy, which includes surgery, radiation therapy, and chemotherapy with temozolomide, the median survival is only 14.6 months. Once patients fail temozolomide, there are no other proven therapies, although other chemotherapies, bevacizumab, and tyrosine kinase inhibitors are often tried. Because tumors are different between patients, outcomes vary among patients. For example, temozolomide, though recommended to all patients with GBM as the only chemotherapy to improve survival, is also known not to be effective in patients with o6-methylguanine-DNA-methyltransferase (MGMT) unmethylated tumors. This example underscores the idea that if each tumor is different, and that perhaps there would be better outcomes if each tumor was treated uniquely.

Genomic sequencing is a technology that can be employed to identify specific characteristics of each tumor as compared to healthy cells. Since 2008, genomic sequencing technology has advanced significantly, having entered the era of next generation sequencing, and simultaneously, the cost of using this technology has dramatically decreased, nearing the cost of some currently used diagnostic tests such as MRI. In this study, the investigators plan to assess the usefulness of this technology and its analysis as a method of guiding treatment choices for the individual patient with GBM.

The investigators plan to sequence tumor/normal from GBM patients to identify mutations. The mutations will be analyzed for potential drug targets for treatment and recommendations for treatment will be suggested if any are identified. If the clinician implements the recommendations, clinical follow up data will be collected. The investigators will compare clinical outcomes, such as survival to historical controls undergoing standard of care treatment to assess whether this genomic guided, individualized therapy determination improves these measures.

In addition, the investigators plan to use next generation sequencing methods to determine whether the presence of brain messenger ribonucleic acid (mRNA) and miRNA can be detected in the peripheral blood and whether there is biological relevance to their presence if detected.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma multiforme
* Enough tumor tissue available from initial surgery to obtain at least 5 ug DNA and 5 ug RNA
* Sufficient blood sample to obtain 5 ug DNA and 5 ug RNA
* Karnofsky score at least 60
* Life expectancy at least 6 months

Exclusion Criteria:

* Subjects not interested in further treatment of their brain tumor

Ages: 3 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with glioblastoma
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-03-12 (Actual); Primary Completion 2017-07-07 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Identification of targetable variants in the tumor | 6 months
  Identification of variants in each tumor that are potential drug targets

CONTACTS AND LOCATIONS:
Overall Officials: Robert Darnell, MD, PhD, Principal Investigator — Rockefeller University
Locations (7):
- United States (7):
  - New York University Langone Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Rockefeller University, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Lenox Hill Hospital, New York, New York
  - North Shore University Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
The data will be coded and shared with members of the collaboration.

REFERENCES:
- [Background] Gormally E, Caboux E, Vineis P, Hainaut P. Circulating free DNA in plasma or serum as biomarker of carcinogenesis: practical aspects and biological significance. Mutat Res. 2007 May-Jun;635(2-3):105-117. doi: 10.1016/j.mrrev.2006.11.002. Epub 2007 Jan 25. PMID 17257890
- [Background] Hegi ME, Diserens AC, Godard S, Dietrich PY, Regli L, Ostermann S, Otten P, Van Melle G, de Tribolet N, Stupp R. Clinical trial substantiates the predictive value of O-6-methylguanine-DNA methyltransferase promoter methylation in glioblastoma patients treated with temozolomide. Clin Cancer Res. 2004 Mar 15;10(6):1871-4. doi: 10.1158/1078-0432.ccr-03-0384. PMID 15041700
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Derived] Wrzeszczynski KO, Frank MO, Koyama T, Rhrissorrakrai K, Robine N, Utro F, Emde AK, Chen BJ, Arora K, Shah M, Vacic V, Norel R, Bilal E, Bergmann EA, Moore Vogel JL, Bruce JN, Lassman AB, Canoll P, Grommes C, Harvey S, Parida L, Michelini VV, Zody MC, Jobanputra V, Royyuru AK, Darnell RB. Comparing sequencing assays and human-machine analyses in actionable genomics for glioblastoma. Neurol Genet. 2017 Jul 11;3(4):e164. doi: 10.1212/NXG.0000000000000164. eCollection 2017 Aug. PMID 28740869
- See also: Wetterstrand KA. DNA Sequencing Costs: Data from the NHGRI Genome SequencingProgram (GSP) — http://www.genome.gov/sequencingcosts